CLINICAL TRIAL: NCT02388646
Title: Energy Dispersive Bracing for Conservative Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FRKDJO-RWB-15
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Knee Osteoarthritis; Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis | interventions — Braces; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise Only (Active Comparator): Home exercise program.
  Interventions: Other: Exercise Only
- Brace Only (Active Comparator): Reaction Web brace.
  Interventions: Device: Brace Only
- Bracing + Exercises (Active Comparator): Reaction Web brace and home exercises.
  Interventions: Other: Bracing + Exercises

INTERVENTIONS:
Other: Exercise Only — This group will be given a set of 2 exercises to complete at home. The exercises are designed to strengthen the quadriceps muscle group.
  Arms: Exercise Only
Device: Brace Only — This group will be fitted with a Reaction Web brace and asked to wear it when going about activities of daily living.
  Arms: Brace Only
Other: Bracing + Exercises — This group will be asked to both wear the Reaction Web brace during activities of daily living and complete a set of 2 exercises designed to strengthen the quadriceps muscle group.
  Arms: Bracing + Exercises

SUMMARY:
The goal of this study is to explore the effectiveness of a commercially available, over-the-counter knee brace in the conservative treatment of knee osteoarthritis. Participants will either be fitted with a brace and told to wear it every day during normal activities, fitted with the brace and given instructions on a set of quadriceps strengthening exercises to complete twice daily, every day, or be given the exercise instructions, but not fitted with a brace. Functional and subjective outcomes will be collected preoperatively and at 6 and 12 weeks from baseline, with the goal of informing the effectiveness of bracing alone versus a home exercise program, and whether the combination of those provides the most therapeutic benefit to participants.

ELIGIBILITY:
Inclusion Criteria:

* Subject is being treated for knee joint pain
* Subject is willing and able to comply with the evaluation schedule

Exclusion Criteria:

* Subject is undergoing surgery during the follow-up window that would limit their ability to comply with the evaluation schedule and/or significantly affect the outcomes measures
* Subject has current alcohol, opioid, or other drug dependence
* Subject is taking prescribed medication for pain other than in the knee joint (e.g. back pain)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Kolisek, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- OrthoIndy, Greenwood, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, only averages and summaries where all participant data is combined.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise Only | Brace Only | Bracing + Exercises
Started | 20 | 20 | 20
Completed | 16 | 19 | 14
Not Completed | 4 | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Only | Brace Only | Bracing + Exercises | Total
Number analyzed (Participants) | 16 | 19 | 14 | 49
Age, Continuous [Mean (Full Range); unit: years] | 67 [56 to 76] | 64 [50 to 76] | 66 [51 to 78] | 66 [50 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 6 | 21
  Male | 9 | 11 | 8 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Laterality [Count of Participants; unit: Participants]
  Right | 8 | 9 | 7 | 24
  Left | 8 | 10 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Pain Using the Visual Analog Scale
Description: The Visual Analog Scale (VAS) consists of a 100mm horizontal line with the words "No Pain" (score of 0) and "Pain as bad as it could possibly be" (score of 100) written on opposite ends. Participants will be asked to mark on the line where their pain is in relation to the two extremes. Measurement is taken from the left-hand side of the line to the mark and reported as a score out of 100. The difference between the baseline score and score at the 3-month study visit was compared between study arms.
Time Frame: Baseline and 3-month Visit
Population: Change from baseline reported in table
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Exercise Only | Brace Only | Bracing + Exercises
Number analyzed (Participants) | 16 | 19 | 14
score on a scale
  Baseline Average VAS Pain Score | 48.7 [4.0 to 97.0] | 62.6 [17.0 to 98.0] | 50.8 [2.0 to 92.0]
  3-Month Average VAS Pain Score | 27.1 [3.5 to 62.0] | 20.7 [1.0 to 48.0] | 13.2 [0.0 to 75.0]

2. Secondary Outcome: Change in Quadriceps Force
Description: Change in quadriceps force is the difference between average quadriceps force measurements (in Newtons) obtained at the 3-month postoperative follow-up minus the average quadriceps force measurement at baseline. Averages are stratified by study arm. Negative values indicate a reduction in quadriceps force from baseline to 3-month.
Time Frame: Baseline and 3-month Visit
Population: Normalized quadriceps force values reported in data table by study arm.
Measure: Mean (Full Range); unit: Newtons (N)
Arm/Group | Exercise Only | Brace Only | Bracing + Exercises
Number analyzed (Participants) | 16 | 19 | 14
Newtons (N) | .25 [-4.65 to 1.33] | .15 [-3.37 to 1.42] | .31 [-3.33 to 1.80]

ADVERSE EVENTS:
Arm/Group | Exercise Only | Brace Only | Bracing + Exercises
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/19 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No